CLINICAL TRIAL: NCT04021381
Title: Citrate Salts for Stone-free Result After Flexible Ureterorenoscopy for Inferior Calyx Calculi: a Randomized Placebo Controlled Trial
Brief Title: Citrate Salts for Stone-free Result After Flexible Ureterorenoscopy for Inferior Calyx Calculi
Acronym: CiRUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P170933J; 2018-A03500-55 (Other: ANSM)
Record Dates: First submitted 2019-05-24; First posted 2019-07-16 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Urolithiasis; Calyx; Calculus
Keywords: Urolithiasis; Urinary Calculi; Ureteroscopy; Residual fragments; Morphoconstitutional analysis; Citrate
MeSH Terms: conditions — Urolithiasis; Calculi; Urinary Calculi | interventions — potassium-magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium and magnesium citrate (Experimental): Patients are treated with potassium and magnesium citrate
  Interventions: Dietary Supplement: Potassium and magnesium citrate
- Placebo (Placebo Comparator): Patients are treated with placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Potassium and magnesium citrate — Patients are treated with potassium and magnesium citrate 5.2 grams daily during 3 months, following flexible ureterorenoscopy for inferior calyx urolithiasis.
  Other Names: Lithos
  Arms: Potassium and magnesium citrate
Dietary Supplement: Placebo — Patient are treated with placebo 5.2 grams daily during 3 months, following flexible ureterorenoscopy for inferior calyx urolithiasis.
  Arms: Placebo

SUMMARY:
The prevalence of urolithiasis is around 10 % in the French population. It is thus a major public health issue. When the stone is not spontaneously removed, interventions such as extracorporeal lithotripsy or flexible ureteroscopy (F-URS) are performed. F-URS is usually preferred in renal stones > 7 mm in comparison with lithotripsy, with better results. Efficacy of ureteroscopy is based on the "stone-free rate" (SFR) at 3 months. A SFR index is assessed according to the existence of residual fragments and their size. SFR score 1 (fragment ≤ 1mm) has been poorly studied, and is supposed to occur in 60% of cases. These residual fragments account for the high frequency of recurrence, probably favored by crystals aggregation and growth of these fragments under supersaturated urines.

Indeed, calcium stones risk factors are urine supersaturation and crystal growth inhibitors deficiency. Citrate is the major crystal growth inhibitor in human urine. A hypocitraturia is reported in half of the lithiasic population.

Consequently, citrate salts appear as an interesting therapeutic option, in order to slow crystal growth but also to chelate calcium, and consequently to solubilize stones in situ. However, to date, there is no available controlled study after surgical intervention such as flexible ureteroscopy.

The aim of the investigator's study is to evaluate the efficacy of a 3-month potassium and magnesium citrate treatment following ureteroscopy on the elimination of residual fragments (SFR score 1).

DETAILED DESCRIPTION:
The screening visit takes place 3 months to 3 days before the baseline visit. Patient will be informed of the study protocol by the surgeon who will perform the flexible ureteroscopy. As usual in clinical practice, a CT scan will be routinely performed. CT-scan interpretation will be centralized and performed blindly.

At the ureteroscopy day (baseline visit: Some sites, according to their usual practice, may admit their patients to hospital the day before the surgery (D-1)), inclusion and exclusion criteria will be checked by the surgeon. A second information on the study protocol will be given and the protocol consent will be signed.

The day of hospital admission, blood and urine will be collected by a nurse in order to define stone risk factors and other comorbidities after informed consent of the patients. Then patients will undergo ureteroscopy.

Stone fragments will be sent for analysis to the stone centre Laboratory (Tenon Hospital, Paris) with images of the stones during surgery (morphoconstitutional analysis).

Patients will be randomized for treatment within 7 days following F-URS, and after verification of randomization criteria. If the randomisation criteria are not completed, the patient will end its participation to the study.

Else, the patient is randomized and treatment for 3 months (placebo or citrate salts, blinded) will be delivered by the investigational site and administration will begin the day following surgery, thus discharge. A 33 cl glass will be provided for the administration of the treatment. Furthermore 24-hour urine collection will be explained and patients will be given the vessel in order to collect urine at M3 visit.

The end of study visit will take place at 3 months +/- 10 days after ureteroscopy visit.

Medical check-up by the urologist in charge, including a CT-scan and blood and urine biological tests under randomized treatment.

Randomized treatment will be stopped the day of this M3 visit. Adverse events (including drug tolerance, urinary symptoms) and date of stent removal if any will be collected. Compliance will be assessed, using a log book.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Efficient contraceptive method in women of childbearing age
* At least one renal urolithiasis 10 ≤ size ≤ 20 mm
* No recent ureterorenoscopy (< 6 months)
* Planned flexible ureterorenoscopy procedure with holmium-laser dusting
* CT-scan performed within 3 months before surgery
* Affiliation to a social security regime
* Informed consent

Exclusion Criteria:

* Stone density < 700 UH on pre-operative CT-scan
* History of infectious renal stones or monogenic lithiasic disease (cystinuria, primary hyperoxaluria)
* Obstructive urinary tract malformation Cacchi-Ricci disease, Horseshoe kidney
* Chronic renal failure (eGFR<30 ml/min/1.73m²)
* Ongoing renal colic (within 7 days)
* Untreated urinary tract infection (within 7 days)
* Contraindications to ureterorenoscopy: coagulation disorders, high anesthetic risk
* Contraindications to potassium and magnesium citrate: known hyperkalemia, known hypermagnesemia, uncontrolled diabetes, acute dehydration
* Pregnant or breastfeeding women
* Patient deprived of liberty or under legal protection measure (tutorship or curatorship);
* Participation in another therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Stone-free result | 3 months
  Percentage of stone-free patients (SFR score 0 and 1) between the 2 groups at 3 months after ureteroscopy assessed by non-injected, low irradiation, thin slice CT-scan.

SECONDARY OUTCOMES:
SFR score 2, 3 and 4 | 3 months
  Percentage of SFR score 2, 3 and 4 in the 2 groups at 3 months assessed by non-injected, low irradiation, thin slice CT-scan
Urine supersaturation index | 3 months
  Urine supersaturation index calculation based on the combination of urine pH, calciuria, phosphaturia, uricosuria, oxaluria) at 3 months in the two groups
To evaluate the Safety of potassium and magnesium citrate: Percentage of patients with at least one adverse event throughout the study | 3 months
  Percentage of patients with at least one adverse event throughout the study and collected at 3 months: epigastralgia, nausea, vomiting, bloating, constipation, diarrhea and urinary tract infection.
  Mean USSQ (ureteral stone symptom questionnaire) score in each group.
To evaluate the compliance of potassium and magnesium citrate as assessed by citraturia | 3 months
  24-hour and fasting citraturia (mmol/L) at 3 months.
To evaluate the compliance of potassium and magnesium citrate as assessed by urinary pH | 3 months
  24-hour and fasting pH at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie TABIBZADEH, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department : Exploration fonctionnelles rénales, Centre de la lithiase Hôpital TENON, Paris, France

IPD SHARING:
Plan to Share IPD: No